CLINICAL TRIAL: NCT03365882
Title: S1613, A Randomized Phase II Study of Trastuzumab and Pertuzumab (TP) Compared to Cetuximab and Irinotecan (CETIRI) in Advanced/Metastatic Colorectal Cancer (mCRC) With HER-2 Amplification
Brief Title: S1613, Trastuzumab and Pertuzumab or Cetuximab and Irinotecan Hydrochloride in Treating Patients With Locally Advanced or Metastatic HER2/Neu Amplified Colorectal Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1613; NCI-2016-01422 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1613; S1613 (Other: SWOG); S1613 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2017-10-02; First posted 2017-12-07 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Colon Adenocarcinoma; ERBB2 Gene Amplification; Rectal Adenocarcinoma; Recurrent Colon Carcinoma; Recurrent Rectal Carcinoma; Stage III Colon Cancer AJCC v7; Stage III Rectal Cancer AJCC v7; Stage IIIA Colon Cancer AJCC v7; Stage IIIA Rectal Cancer AJCC v7; Stage IIIB Colon Cancer AJCC v7; Stage IIIB Rectal Cancer AJCC v7; Stage IIIC Colon Cancer AJCC v7; Stage IIIC Rectal Cancer AJCC v7; Stage IV Colon Cancer AJCC v7; Stage IV Rectal Cancer AJCC v7; Stage IVA Colon Cancer AJCC v7; Stage IVA Rectal Cancer AJCC v7; Stage IVB Colon Cancer AJCC v7; Stage IVB Rectal Cancer AJCC v7
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Irinotecan; pertuzumab; 2C4 antibody; Trastuzumab; PF-05280014

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm I (pertuzumab, trastuzumab) (Experimental): Patients receive pertuzumab IV over 30-60 minutes and trastuzumab IV over 30-120 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pertuzumab; Biological: Trastuzumab; Device: HER-2 testing
- Arm II (cetuximab, irinotecan hydrochloride) (Experimental): Patients receive cetuximab IV over 60-120 minutes and irinotecan hydrochloride IV over 90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients with documented disease progression may optionally crossover to Arm I.
  Interventions: Biological: Cetuximab; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Device: HER-2 testing

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm II (cetuximab, irinotecan hydrochloride)
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E
  Arms: Arm II (cetuximab, irinotecan hydrochloride)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pertuzumab — Given IV
  Other Names: 2C4; 2C4 Antibody; MoAb 2C4; Monoclonal Antibody 2C4; Perjeta; rhuMAb2C4; RO4368451
  Arms: Arm I (pertuzumab, trastuzumab)
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar PF-05280014
  Arms: Arm I (pertuzumab, trastuzumab)
Device: HER-2 testing — Central testing of HER-2 for eligibility

SUMMARY:
This randomized phase II trial studies how well trastuzumab and pertuzumab work compared to cetuximab and irinotecan hydrochloride in treating patients with HER2/neu amplified colorectal cancer that has spread from where it started to other places in the body and cannot be removed by surgery. Monoclonal antibodies, such as trastuzumab and pertuzumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as cetuximab and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving trastuzumab and pertuzumab may work better compared to cetuximab and irinotecan hydrochloride in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of trastuzumab and pertuzumab (TP) (Arm 1) in HER-2 amplified metastatic colorectal cancer (mCRC) by comparing progression-free survival (PFS) on TP compared to control arm (Arm 2) of cetuximab and irinotecan hydrochloride (irinotecan) (CETIRI).

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate (ORR), including confirmed complete and partial response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, in treatment Arms 1 and 2.

II. To evaluate the overall survival (OS) in treatment Arms 1 and 2. III. To evaluate the safety and toxicity of TP compared to CETIRI.

TERTIARY OBJECTIVES:

I. To estimate the rates of PFS, OS, and ORR in patients who crossover to TP (Arm 3) after disease progression on CETIRI.

II. To bank images for future retrospective analysis. III. To evaluate if HER-2/centromeric probe (CEP17) signal ratio and HER-2 gene copy number (GCN) are predictive of clinical efficacy for patients receiving TP versus CETIRI.

IV. To bank tissue and blood samples for other future correlative studies from patients enrolled on the study.

OUTLINE: Patients with HER2 gene amplification are randomized to 1 of 2 arms.

ARM I: Patients receive pertuzumab intravenously (IV) over 30-60 minutes and trastuzumab IV over 30-120 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive cetuximab IV over 60-120 minutes and irinotecan hydrochloride IV over 90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients with documented disease progression may optionally crossover to Arm I.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 INITIAL REGISTRATION: HER2 TESTING
* Patients must have histologically or cytologically documented adenocarcinoma of the colon or rectum that is metastatic or locally advanced and unresectable
* Mutation results:

  * All patients must have molecular testing performed in a Clinical Laboratory Improvement Act (CLIA) certified lab which includes which includes KRAS and NRAS gene and exon 15 of BRAF gene (BRAF V600E mutation); patients with any known activating mutation in exon 2 [codons 12 and 13], exon 3 [codons 59 and 61] and exon 4 [codons 117 and 146]) of KRAS/NRAS genes and in exon 15 (BRAFV600E mutation) of BRAF gene are not eligible
* Patients must not have been treated with any of the following prior to step 1 initial registration:

  * Cetuximab, panitumumab, or any other monoclonal antibody against EGFR or inhibitor of EGFR
  * HER-2 targeting for treatment of colorectal cancer; patients who have received prior trastuzumab or pertuzumab for other indications such as prior history of adjuvant or neoadjuvant breast cancer treatment prior to the development of advanced colorectal cancer are eligible
* Patients must not have had history of severe toxicity and intolerance to or hypersensitivity to irinotecan or any other study drug; patients must not have had a severe infusion-related reaction during any prior therapy with pertuzumab or trastuzumab
* Patients must have tumor slides available for submission for HER-2 testing; HER-2 testing must be completed by the central lab prior to step 2 randomization
* Patients must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines; for step 1 initial registration, the appropriate consent form is the step 1 consent form
* As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* STEP 2 RANDOMIZATION
* Patients must have HER-2 amplification as determined by central testing (3+ or 2+ by immunohistochemistry and HER-2 gene amplification by in situ hybridization with a ratio of HER-2 gene signals to centromere 17 signals >= 2.0)
* Patients must have measurable disease that is metastatic or locally advanced and unresectable; imaging used to assess all disease per RECIST 1.1 must have been completed within 28 days prior to step 2 randomization; all disease must be assessed and documented on the Baseline Tumor Assessment Form
* Patients must have had at least one prior regimen of systemic chemotherapy for metastatic or locally advanced, unresectable disease; patients must have progressed following the most recent therapy; prior treatment with irinotecan is allowed; for patients that received adjuvant chemotherapy: prior treatment for metastatic disease is not required for patient who experienced disease recurrence during or within 6 months of completion of adjuvant chemotherapy; if the patient received one line of adjuvant treatment and had disease recurrence after 6 months of completing chemotherapy, patients will only be eligible after failing one additional line of chemotherapy used to treat the metastatic or locally advanced, unresectable disease; patients who have received >= 3 lines of systemic chemotherapy for metastatic or locally advanced, unresectable disease are not eligible
* Patients must have completed prior chemotherapy, immunotherapy, or radiation therapy at least 14 days prior to step 2 randomization and all toxicity must be resolved to Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0 grade 1 (with the exception of CTCAE v4.0 grade 2 neuropathy) prior to step 2 randomization
* Brain metastases are allowed if they have been adequately treated with radiotherapy or surgery and stable for at least 30 days prior to step 2 randomization; eligible patients must be neurologically asymptomatic and without corticosteroid treatment for at least 7 days prior to step 2 randomization
* Patients must have a Zubrod performance status of 0 or 1
* Patients must have a complete physical examination and medical history within 28 days prior to step 2 randomization
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 75,000/mcL
* Hemoglobin >= 9 g/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both =< 5 x institutional upper limit of normal (IULN)
* Bilirubin =< 1.5 mg/dL
* Calculated creatinine clearance > 30 ml/min within 14 days prior to step 2 randomization
* Patients who have had an echocardiogram performed within 6 months prior to step 2 randomization must have ventricular ejection fraction (left ventricular ejection fraction [LVEF]) >= 50% or >= within normal limits for the institution
* Patients must not have an uncontrolled intercurrent illness including, but not limited to diabetes, hypertension, severe infection, severe malnutrition, unstable angina, class III-IV New York Heart Association (NYHA) congestive heart failure, ventricular arrhythmias, active ischemic heart disease, or myocardial infarction within 6 months prior to step 2 randomization
* Patients must not have any known previous or concurrent condition suggesting susceptibility to hypersensitivity or allergic reactions, including, but not limited to: known hypersensitivity to any of the study treatments or to excipients of recombinant human or humanized antibodies; patients with mild or seasonal allergies may be included after discussion with the study chairs
* Patients must not be planning treatment with other systemic anti-cancer agents (e.g., chemotherapy, hormonal therapy, immunotherapy) or other treatments not part of protocol-specified anti-cancer therapy including concurrent investigational agents of any type
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, ductal carcinoma in situ, other low grade lesions such as incidental appendix carcinoid, or any other cancer from which the patient has been disease and treatment free for two years; prostate cancer patients on active surveillance are eligible
* Patients must not be pregnant or nursing; females of child-bearing potential must have a negative serum pregnancy test within 7 days prior to registration; women/men of reproductive potential must have agreed to use an effective contraceptive method while on study and for at least 7 months after the last dose of study treatment; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must be given the opportunity to consent to the optional submission of tissue for future research
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines; the appropriate consent form for this registration is the step 2 consent form
* STEP 2 RANDOMIZATION: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): Patients must have documented disease progression while on CETIRI (Arm 2) on this protocol; the Follow-up Tumor Assessment Form documenting disease progression must be submitted to Southwest Oncology Group (SWOG) prior to step 3 crossover registration; registration to step 3 crossover must be within 28 days of discontinuation of CETIRI protocol treatment; patients going off treatment for any other reason are not eligible
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): Patients must have a Zubrod performance status of 0 or 1
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): ANC >= 1,500/mcL
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): Platelets >= 75,000/mcL
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): Hemoglobin >= 9 g/dL
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): AST and ALT both =< 5 x institutional upper limit of normal (IULN)
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): Bilirubin =< 1.5 mg/dL
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): Calculated creatinine clearance > 30 ml/min within 14 days prior to step 3 crossover registration
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): Patients must have left ventricular ejection fraction (LVEF) >= 50% or >= lower limit of normal for the institution by echocardiogram within 14 days prior to step 3 crossover registration
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): Patients must have a magnesium, potassium, calcium, sodium, bicarbonate, and chloride performed within 14 days prior to step 3 crossover registration
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines; the appropriate consent form for this registration is the step 2 consent form
* STEP 3 CROSSOVER REGISTRATION (OPTIONAL): As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2025-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanwal Raghav, Principal Investigator — SWOG Cancer Research Network
Locations (798):
- United States (786):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - City of Hope Corona, Corona, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - City of Hope Mission Hills, Mission Hills, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mills Health Center, San Mateo, California
  - City of Hope - Santa Clarita, Santa Clarita, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope Upland, Upland, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - City of Hope West Covina, West Covina, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center - Guiford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Low Country Cancer Care, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Franciscan Saint Elizabeth Health - Lafayette East, Lafayette, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Jennie Edmundson Memorial Hospital, Council Bluffs, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Bloomfield, Bloomfield, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Levine Cancer Institute - Rutherford, Forest City, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kenansville, Kenansville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Vidant Oncology-Richlands, Richlands, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Johnston Memorial Hospital, Smithfield, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Bryn Mawr Health Center, Newtown Square, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Kent Hospital, Warwick, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Scott and White Healthcare Round Rock, Round Rock, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Puerto Rico (12):
  - Advance Oncology Center, Aguadilla
  - Doctor's Cancer Center-Arecibo, Arecibo
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Hematologia Oncologia San Pablo, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Primary Care Physician Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan
  - Centro de Hematologia y Oncologia del Sur, Santa Isabel

REFERENCES:
- [Derived] Raghav KPS, Guthrie KA, Tan B Jr, Denlinger CS, Fakih M, Overman MJ, Dasari NA, Corum LR, Hicks LG, Patel MS, Esparaz BT, Kazmi SM, Alluri N, Colby S, Gholami S, Gold PJ, Chiorean EG, Kopetz S, Hochster HS, Philip PA. Trastuzumab Plus Pertuzumab Versus Cetuximab Plus Irinotecan in Patients With RAS/BRAF Wild-Type, HER2-Positive, Metastatic Colorectal Cancer (S1613): A Randomized Phase II Trial. J Clin Oncol. 2025 Apr 10;43(11):1348-1357. doi: 10.1200/JCO-24-01710. Epub 2025 Jan 6. PMID 39761503

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 240 participants were screened for HER-2 amplification, 54 participant were HER-2 positive and randomized to therapy, 1 patient is not analyzable due to withdrawal of consent and refusal of protocol treatment.
Groups:
- Trastuzumab + Pertuzumab: Participants receive pertuzumab intravenously (IV) over 30-60 minutes and trastuzumab IV over 30-120 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Cetuximab + Irinotecan: Participants receive cetuximab IV over 60-120 minutes and irinotecan hydrochloride IV over 90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Participants with documented disease progression may optionally crossover to Arm I.
Period: Randomization
Arm/Group | Trastuzumab + Pertuzumab | Cetuximab + Irinotecan
Started | 26 | 28
Progressed and Crossed Over | 0 | 20
Completed | 0 | 20
Not Completed | 26 | 8
Not completed — Still Receiving Protocol Treatment | 2 | 0
Not completed — Adverse Event | 1 | 2
Not completed — Refusal Unrelated to Adverse Event | 0 | 1
Not completed — Progression/Relapse | 21 | 3
Not completed — Death | 1 | 0
Not completed — Other - Not Protocol Specified | 1 | 1
Not completed — Major Protocol Deviation | 0 | 1
Period: Crossover: Trastuzumab + Pertuzumab
Arm/Group | Trastuzumab + Pertuzumab | Cetuximab + Irinotecan
Started | 0 | 20
Completed | 0 | 0
Not Completed | 0 | 20
Not completed — Still Receiving Protocol Treatment | 0 | 1
Not completed — Progression/Relapse | 0 | 13
Not completed — Other - Not Protocol Specified | 0 | 4
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab + Pertuzumab | Cetuximab + Irinotecan | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Median (Full Range); unit: years] | 56.2 [32.1 to 83.8] | 59.1 [38.9 to 75.2] | 57.6 [32.1 to 83.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic: Yes | 1 | 2 | 3
  Hispanic: No | 23 | 25 | 48
  Hispanic: Unknown | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 19 | 21 | 40
  Race: Black | 1 | 4 | 5
  Race: Asian | 4 | 1 | 5
  Race: Unknown | 2 | 1 | 3
Number of Participants with Prior Use of Irinotecan [Count of Participants; unit: Participants]
  Yes | 11 | 13 | 24
  No | 15 | 14 | 29
HER2/CEP17 Ratio [Count of Participants; unit: Participants]
  >5 | 19 | 20 | 39
  <=5 | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival(PFS)
Description: To evaluate the efficacy of trastuzumab and pertuzumab (TP) in HER-2 amplified metastatic colorectal cancer (mCRC) by comparing progression-free survival (PFS) on TP compared to control arm of cetuximab and irinotecan (CETIRI). Progression-free survival is defined as the time from date of randomization to date of first documentation of progression. Using RECIST 1.1, progression is defined as a 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed and an absolute increase of at least 0.5 cm, unequivocal progression of non-measurable disease in the opinion of the treating physician, appearance of any new lesion/site, death due to disease without prior documentation of progression and without symptomatic deterioration (defined as, global deterioration of health status requiring discontinuation of treatment without objective evidence of progression), or death due to any cause.
Time Frame: Up to 3 years post randomization
Population: This population includes the 53 eligible and evaluable participants. 26 in the Trastuzumab + Pertuzumab arm and 27 in the Cetuximab + Irinotecan arm.
Measure: Median (Full Range); unit: Months
Arm/Group | Trastuzumab + Pertuzumab | Cetuximab + Irinotecan
Number analyzed (Participants) | 26 | 27
Months | 4.7 [1.9 to 7.6] | 3.7 [1.6 to 6.7]
Statistical Analysis 1: Comparison: Trastuzumab + Pertuzumab vs Cetuximab + Irinotecan; Test type: Superiority; p = 0.44, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.43 to 1.45]

2. Secondary Outcome: Overall Response Rate (ORR) for TP and CETIRI Treatment Arms
Description: To evaluate the overall response rate (ORR), including confirmed complete and partial response per RECIST 1.1, in the TP and CETIRI treatment arms. Overall response rate includes complete response(CR) and partial response(PR). Complete response is defined as complete disappearance of all target and non-target lesions and no related symptoms. Partial response is defined as a greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions for patients with at least one measurable lesion.
Time Frame: From baseline, through duration of treatment (once per cycle while on treatment), and every 8 weeks after treatment until progression, up to 3 years after the last accrual to registration step 2
Population: This population includes the 53 eligible and evaluable participants. 26 participants in the Trastuzumab + Pertuzumab arm and 27 participants in the Cetuximab + Irinotecan arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab + Pertuzumab | Cetuximab + Irinotecan
Number analyzed (Participants) | 26 | 27
Participants | 9 | 7

3. Secondary Outcome: 2 Year Overall Survival (OS) for TP and CETIRI Treatment Arms
Description: Percentage of participants still alive 2 years after the last accrual to registration step 2. Overall survival is defined as time from date of registration to date of death due to any cause. Patients last known to be alive are censored at their last contact date.
Time Frame: from the date of the last accrual to registration step 2 to date of death due to any cause, up to 2 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab + Pertuzumab | Cetuximab + Irinotecan
Number analyzed (Participants) | 26 | 27
percentage of participants | 67.1 [44.6 to 82.1] | 56.7 [35.2 to 73.5]
Statistical Analysis 1: Comparison: Trastuzumab + Pertuzumab vs Cetuximab + Irinotecan; Test type: Superiority; p = 0.17, Log Rank

4. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs.
Description: Routine toxicities were evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0, and SAEs were evaluated according to CTCAE version 5.0. Only adverse events that are possibly, probably, or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow-up until death or 3 years post Step 2 Randomization.
Population: Participants who were eligible and received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Arm/Group | Trastuzumab + Pertuzumab | Cetuximab + Irinotecan
Number analyzed (Participants) | 26 | 26
Participants
  Abdominal pain | 1 | 0
  Alanine aminotransferase increased | 1 | 0
  Alkaline phosphatase increased | 1 | 0
  Anemia | 0 | 1
  Anorexia | 0 | 1
  Atrial fibrillation | 1 | 0
  Diarrhea | 0 | 2
  Dyspnea | 1 | 0
  Fatigue | 0 | 2
  Gastrointestinal disorders - Other, specify | 0 | 2
  Hypokalemia | 0 | 1
  Hypomagnesemia | 0 | 1
  Infusion related reaction | 1 | 0
  Leukocytosis | 0 | 1
  Lymphocyte count decreased | 1 | 0
  Rash acneiform | 0 | 3
  Rash maculo-papular | 1 | 2
  Thromboembolic event | 0 | 1
  Vomiting | 1 | 1

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post Step 2 Randomization.
Description: CTCAE version 5.0 was used for reporting SAEs and CTCAE version 4.0 was used for routine toxicity reporting. All-Cause mortality was assessed in all analyzable participants, 26 participants in the Trastuzumab + Pertuzumab arm and 27 participants in the Cetuximab + Irinotecan arm. Due to 1 participant refusal of treatment, there were only 26 participants in the Cetuximab + Irinotecan arm that were evaluable for AEs and 26 participants in the Trastuzumab + Pertuzumab arm evaluable for AEs.
Groups:
- Cetuximab + Irinotecan: Participants receive cetuximab IV over 60-120 minutes and irinotecan hydrochloride IV over 90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Participants with documented disease progression may optionally crossover to Arm I. The number of affected participants in All-Cause Mortality includes participants that died after they crossed over to Arm I.
- Crossover: Trastuz +Pertuz: Following radiographic documentation by RECIST 1.1 of disease progression, participants initially randomized and treated with Cetuximab + Irinotecan may register to Step 3 Crossover Registration to be treated with Trastuzumab + Pertuzumab according to Arm/Group 1's description.
Arm/Group | Trastuzumab + Pertuzumab | Cetuximab + Irinotecan | Crossover: Trastuz +Pertuz
All-Cause Mortality (participants affected / at risk) | 9/26 | 18/27 | 12/20
Serious Adverse Events (participants affected / at risk) | 8/26 | 1/26 | 5/20
Other Adverse Events (participants affected / at risk) | 23/26 | 26/26 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Pertuzumab (N=26) | Cetuximab + Irinotecan (N=26) | Crossover: Trastuz +Pertuz (N=20)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Infusion related reaction (General disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 0 | 0 | 1
Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Pertuzumab (N=26) | Cetuximab + Irinotecan (N=26) | Crossover: Trastuz +Pertuz (N=20)
Anemia (Blood and lymphatic system disorders) | 4 | 8 | 3
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 3 | 0
Blurred vision (Eye disorders) | 0 | 0 | 1
Eye disorders-Other (Eye disorders) | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 6 | 1
Ascites (Gastrointestinal disorders) | 0 | 2 | 0
Bloating (Gastrointestinal disorders) | 0 | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 8 | 3
Diarrhea (Gastrointestinal disorders) | 15 | 14 | 11
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 3 | 2
Mucositis oral (Gastrointestinal disorders) | 4 | 5 | 2
Nausea (Gastrointestinal disorders) | 5 | 13 | 4
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 6 | 0
Chills (General disorders) | 4 | 0 | 3
Edema limbs (General disorders) | 4 | 1 | 2
Fatigue (General disorders) | 9 | 14 | 10
Fever (General disorders) | 1 | 0 | 1
Flu like symptoms (General disorders) | 2 | 2 | 1
General disorders and admin site conditions - Other (General disorders) | 1 | 0 | 1
Infusion related reaction (General disorders) | 1 | 3 | 3
Irritability (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 1
Pain (General disorders) | 3 | 2 | 2
Infections and infestations-Other (Infections and infestations) | 2 | 2 | 0
Paronychia (Infections and infestations) | 0 | 1 | 2
Upper respiratory infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0
Alanine aminotransferase increased (Investigations) | 4 | 4 | 3
Alkaline phosphatase increased (Investigations) | 6 | 5 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 5 | 3
Blood bilirubin increased (Investigations) | 2 | 2 | 0
Creatinine increased (Investigations) | 2 | 0 | 2
Ejection fraction decreased (Investigations) | 2 | 0 | 0
Investigations-Other (Investigations) | 3 | 2 | 0
Lymphocyte count decreased (Investigations) | 6 | 4 | 2
Neutrophil count decreased (Investigations) | 2 | 5 | 0
Platelet count decreased (Investigations) | 1 | 3 | 2
Weight loss (Investigations) | 0 | 2 | 3
White blood cell decreased (Investigations) | 2 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 6 | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 4 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 7 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 10 | 2
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 4 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 3 | 3
Syncope (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 2 | 1
Hematuria (Renal and urinary disorders) | 1 | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 4 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 10 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 12 | 7
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Hypertension (Vascular disorders) | 3 | 6 | 3
Hypotension (Vascular disorders) | 0 | 2 | 0
Thromboembolic event (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT03365882/Prot_SAP_000.pdf